CLINICAL TRIAL: NCT05117801
Title: Evaluation of Pétale® (Small Hearing Test Equipment for Children) for the Screening of Hearing Disorders in Children From 9 Months to 3 Years Old by the General Practitioner or Pediatrician
Acronym: PETALE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-A02005-52
Record Dates: First submitted 2021-10-28; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Petale; Hearing Disorders; Child Development
MeSH Terms: conditions — Hearing Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children at the general practitioner or pediatrician (Experimental): Children between 9 months and 3 years-old coming to their doctor for any consultation
  Interventions: Device: Petale

INTERVENTIONS:
Device: Petale — The child sits on the companion's lap between the two enclosures, and the investigator observes whether or not he is attracted to a familiar calibrated noise coming from one side or the other.

SUMMARY:
The aim of this study is to confirm the value of this new version of Pétale® ((small equipment for testing the child's hearing) in the daily practice of general practitioners or pediatricians for the screening of hearing disorders in very young children.

DETAILED DESCRIPTION:
The research procedure is auditory stimulation using Pétale® (small equipment for testing the child's hearing) based on the "orientation reflex" ("Ewing" test): the child is seated on the companion's knees between the two enclosures and the investigator observes whether or not he is attracted to a familiar calibrated noise coming from one side or the other.

ELIGIBILITY:
Inclusion Criteria:

* Chil, girl or boy between 9 months and 3 years-old
* Child seen in consultation by a general practitioner or a pediatrician whatever the reason for consultation
* Child attached to a beneficiary of a social security scheme
* Signature of informed consent by parents.

Exclusion Criteria:

* Age greater than 3 years and less than 9 months
* Refusal of one or more parents during the consultation
* State of the child which does not allow the screening test to be carried out

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2022-07-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 2 weeks
  Proportion of children with a hearing impairment assessed by the investigator knowing that they were also assessed with a hearing impairment by ENT specialist.
Specificity | 2 weeks
  Proportion of children without hearing impairment assessed by the investigator knowing that they were also assessed without hearing impairment by ENT.
Positive Predictive Value (PPV): | 2 weeks
  Proportion of children with hearing impairment assessed by both investigator and ENT among children with hearing impairment assessed by ENT.
Negative Predictive Value (NPV) | 2 weeks
  Proportion of children without hearing impairment assessed by both investigator and ENT among children without hearing impairment assessed by ENT.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint-Amé, Lambres-lez-Douai, France